CLINICAL TRIAL: NCT00353782
Title: Disease Pathogenesis and Natural History of Lipid Disorders
Brief Title: Causes and Natural History of Dyslipidemias
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030280; 03-H-0280
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-10-14

CONDITIONS: Hypercholesterolemia; Atherosclerosis
Keywords: Triglyceride; Phospholipids; Free and Esterfied Cholesterol; Polydisperse; Lipoprotein Transport System; Natural History
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyslipidemia: Dyslipidemia

SUMMARY:
This study will evaluate people with dyslipidemias - disorders that affect the fat content in the blood. Fats, or lipids, such as cholesterol and triglycerides, are carried in the blood in particles called lipoproteins. These particles are involved in causing blood vessel diseases that can lead to conditions like atherosclerosis (hardening of the arteries) or heart attack. Participants will undergo accepted medical tests and procedures to evaluate their condition. Most of the test results are helpful in making a diagnosis and in guiding treatment.

People with lipid disorders are eligible for this study. Representative types of patients include those with:

* Plasma cholesterol levels greater than 200 mg/dl or less than 120 mg/dl
* Plasma LDL-C levels greater than 130 mg/dl or less than 70 mg/dl
* Plasma HDL-C levels greater than 70 mg/dl or less than 25 mg/dl
* Unusual cholesterol deposits or xanthomas (nodules of lipid deposits on the skin)

Children under 2 years of age are excluded from the study.

Participants will undergo some or all of the following procedures:

- Plasma evaluation. Apolipoproteins (plasma proteins involved in metabolism of cholesterol, triglycerides, phospholipids, and proteins in the blood) and enzymes involved in lipid metabolism are measured.

DETAILED DESCRIPTION:
The lipoprotein transport system is vital to the delivery of the hydrophobic fats that are carried in the aqueous environment of the blood. The lipoprotein particles that comprise this system are polydisperse and contain triglycerides, free and esterified cholesterol, phospholipids and proteins. Inborn errors in the lipoprotein transport system lead to alterations in both the steady state concentrations of the various lipoproteins and in the metabolism of these particles. These inborn errors lead to both hyperlipoproteinemia and hypolipoproteinemia. Profound changes in the ambient lipoprotein concentrations have a variety of clinical manifestations. The present study protocol is designed to permit a full plasma evaluation of the lipids, lipoproteins and apolipoproteins, in patients with potential genetic defects in these processes. We will use a variety of research plasma assays. These specialized plasma assays are necessary to correctly diagnose and treat patients that present with the more unusual disorders of lipid metabolism; these patients cannot be diagnosed by standard, CLIA- Certified assays and may require tissue or blood cells for diagnosis and adequate treatment. The study population will include patients which are referred to the Lipid Service, Cardiovascular Branch, NHLBI from private care providers, academic institutions or the NHLBI-MDB website, with any of the following potential lipid abnormalities or clinical stigmata associated with dyslipoproteinemias: a) increased plasma levels of cholesterol, triglycerides, HDL-cholesterol or LDL-cholesterol b) decreased plasma concentrations of cholesterol and HDL-cholesterol c) postprandial hyperlipidemia or d) eruptive xanthomas, xanthelasma, tuberous or tendinous xanthomas, or corneal opacities.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Children >= 2 years of age and >12 kg and adults
* Dyslipidemia subjects of interest the group

The following is a representative list of the types of patient presentations with dyslipidemia and potential diagnoses eligible for this protocol:

* Plasma cholesterol levels >200 mg/dl or <120 mg/dl includes patients with diagnoses such as familial hypercholesterolemia, familial combined hyperlipidemia, sitosterolemia, lipoprotein lipase, hepatic lipase or apo-CII deficiency, and dysbetalipoproteinemia.
* Plasma LDL-C levels >130 mg/dl or <70 mg/dl includes patients with diagnoses such as familial hypercholesterolemia, PCSK9, apo3500, familial combined hyperlipidemia, sitosterolemia, dysbetalipoproteinemia, abetalipoproteinemia and hypobetalipoproteinemia.
* Plasma HDL-C levels >70 mg/dl or <25 mg/dl includes patients with deficiency of cholesteryl ester transfer protein, lecithin cholesterol acyltransferase, phospholipid transfer protein, lipoprotein lipase, hepatic lipase, or apo-CII, ANGPTL3, and Tangier disease.
* Plasma triglyceride levels >150 mg/dl includes patients with deficiency of lipoprotein lipase, hepatic lipase or apoC-II, GPIHBP1, LMF1, dysbetalipoproteinemia, Type I, Type IV and Type V hyperlipidemia.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unlimited
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-10-14 (Actual)

PRIMARY OUTCOMES:
permit a full evaluation of the lipoproteins, apolipoproteins, and cellular enzymes and receptors relevant to lipoprotein metabolism in order to accurately diagnose and treat patients with potential genetic defects in these processes | 25 years
  Evaluate Lipids

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Iverius PH, Ostlund-Lindqvist AM. Preparation, characterization, and measurement of lipoprotein lipase. Methods Enzymol. 1986;129:691-704. doi: 10.1016/0076-6879(86)29099-0. No abstract available. PMID 3523161
- [Background] Santamarina-Fojo S, Brewer HB Jr. The familial hyperchylomicronemia syndrome. New insights into underlying genetic defects. JAMA. 1991 Feb 20;265(7):904-8. No abstract available. PMID 1992190
- [Background] Chait A, Iverius PH, Brunzell JD. Lipoprotein lipase secretion by human monocyte-derived macrophages. J Clin Invest. 1982 Feb;69(2):490-3. doi: 10.1172/jci110473. PMID 7056857
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-H-0280.html